CLINICAL TRIAL: NCT05123547
Title: DENTAL CARE OF PATIENTS LIVING WITH HIV, OR COINFECTED HIV / HBV OR HIV / HCV, FOLLOWED IN THE INFECTIOUS DISEASES DEPARTMENT OF CHU CLERMONT-FERRAND
Brief Title: DENTAL CARE OF PATIENTS LIVING WITH HIV
Acronym: DENTA-VIH
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 JACOMET 3; 2021-A01831-40 (Other: 2021-A01831-40)
Record Dates: First submitted 2021-10-18; First posted 2021-11-17 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
Keywords: HIV; Dental care
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is perform to identify oral diseases of people living with HIV (PLWHIV) or co-infected with HBV or HCV.

DETAILED DESCRIPTION:
In the purpose of identifying oral diseases of people living with HIV (PLWHIV) or co-infected with HBV or HCV, we would recruit from 15 10 2021 to 15 04 2022 affiliated to social security scheme PLWHIV adults followed-up in the infectious diseases department of Clermont-Ferrand university hospital who accept participate in order to propose dental individual clinical exams. Anonymous socio-demograpic, medical and dental data will be reported in Redcap. Primary outcomes are the number and type of pathologies identified linked to HIV or not. Statistical analysed will be performed with Stata software. The population will be described by associated numbers and percentages for the categorical variables and by the mean ± standard deviation or median [interquartile interval] for the quantitative variables, with respect to their statistical distribution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient infected with HIV or co-infected with HIV / HBV or HIV / HCV followed in the Infectious Diseases department of Clermont-Ferrand University Hospital and affiliated to a social security scheme.

Exclusion Criteria:

* Minor patient
* Adult patient unable to express his non-opposition to participating in the study or patient who refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people living with HIV
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
description of oral disease linked to HIV or not. | During the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  percentage of patients with oral disease linked to HIV and percentage of patients with oral disease not linked to HIV

SECONDARY OUTCOMES:
Study the factors associated with the presence of oral pathologies linked to HIV. | During the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  bivariate and multivariate analysis of demographic, immunovirologic factors and comorbidities associated to oral diseases linked to HIV
Study the factors associated with the presence of oral pathologies unrelated to HIV. | During the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  bivariate and multivariate analysis of demographic, immunovirologic factors and comorbidities associated with the presence of oral pathologies unrelated to HIV
Compare the prevalence of oral pathologies linked or not to HIV with that found in a previous study carried out in 2003. | During the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  comparison of prevalence of oral diseases in 2021 and those in 2003 in CHU Clermont Ferrand
List the course of dental care of these people during the last 3 years. | During the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  % refusal care, % lost of dental follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christine JACOMET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No